CLINICAL TRIAL: NCT05922813
Title: A Phase I Clinical Trial to Evaluate the Safety and Tolerability of a Single-dose Administration of BMI2004 Inj. (Hyaluronidase, Recombinant) in Healthy Adults
Brief Title: Evaluate the Safety and Tolerability of a Single-dose Administration of BMI2004 Inj.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BMI Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMI2004-SIT-01
Record Dates: First submitted 2023-06-13; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Health, Subjective
Keywords: hyaluronidase; hyaluronidase, recombinant; BMI Korea; BMI2004
MeSH Terms: interventions — Hyaluronoglucosaminidase; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMI2004 Inj. (Experimental): hyaluronidase, recombinant
  Interventions: Biological: BMI2004
- 0.9% NaCl (Placebo Comparator): Normal Saline
  Interventions: Other: 0.9% NaCl

INTERVENTIONS:
Biological: BMI2004 — hyaluronidase, recombinant
  Other Names: hyaluronidase, recombinant
  Arms: BMI2004 Inj.
Other: 0.9% NaCl — Normal Saline
  Arms: 0.9% NaCl

SUMMARY:
A phase I clinical trial to evaluate the safety and tolerability of a single-dose administration of BMI2004 Inj. (hyaluronidase, recombinant) in healthy adults

DETAILED DESCRIPTION:
This study is a phase I clinical trial to evaluate the drug allergic reaction occurring after the single-dose intradermal injection of BMI2004 Inj. and the safety and tolerability after the single-dose subcutaneous injection of BMI2004 in healthy adults. The study consists of Part I and Part II that Part I is the drug allergic reaction evaluation and Part II is the safety evaluation.

Part I (Drug allergic reaction evaluation) : Subjects who provide a written consent to participation in the study will receive the screening test. The subjects determined to be eligible for the study based on the screening test results and inclusion/exclusion criteria are intradermally administered the single-dose test drug (BMI2004 inj.) on the forearm and the single-dose placebo (Dai Han Isotonic Sodium Chloride Inj.) on one the other forearm, respectively, at the baseline visit(Visit 2). Then subjects are investigated for immediate drug allergic reaction occurring within 30 minutes after the administration of the Investigational Products(IPs) and delayed drug allergic reaction occurring between 30 minutes and 48 hours after the administration

Part II (safety evaluation) : Subjects confirmed negative in the drug allergic reaction test at Visit 4 on Part I are randomized either to the single-dose test group (BMI2004 Inj.) or the single-dose placebo group (Dai han Isotonic Sodium Chloride Inj.) at a ratio or 2:1 and subcutaneously administered on the right or left arm.

After the administration of the IPs, the injection site will be monitored. Subjects with no adverse events within 30 minutes after administration may leave while those with adverse events will receive appropriate treatment before leaving. At the follow-up visit(Visit 6 to 8) and the end-of study(EOS) visit (Visit 9), investigation of changes of concomitant medications, safety evaluation, and scheduled assessments are performed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female aged 19 years or above at the screening visit(Visit 1)
2. Female subject who are non-childbearing potential due to menopause or surgery or who have agreed to use methods of contraception during the study, or male subjects with female partners who meet the aforementioned conditions, including º Female subjects who are post-menopausal (Diagnosed with nontherapy-induced amenorrhea or menopause for 12 months or longer) or male subjects with female partners who meet the said conditions º Female subjects who are of non-childbearing potential due to surgery (oophorectomy and/or hysterectomy) or male subjects with female partners who meet the said conditions º Subjects who have agreed to observe absolute sexual abstinence during the study [except for the case of partial sexual abstinence of female subjects (e.g., coitus interruptus in the ovulation or post-ovulation period or the basal body temperature)] º Subjects who have agreed to use the following methods of contraception, if female subjects or female partners of male subjects are women of child-bearing potential (WOCBP) and did not undergo infertility surgery

   - Hormonal contraceptives (implantable form, patch or oral administration)
   * Intrauterine devices(IUD)
   * Double-barrier methods*(Simultaneous use of two of the following methods: Male condoms, female condoms, cervical caps, contraceptive diaphragms, contraceptive sponge, and spermicides) *Simultaneous use of male condoms and female condoms is not considered to be a double barrier method.
3. Subjects with no tattoos, acne, dermatitis, pigmentation, scars, lesions, or damaged skin on the injection site for the investigational products (IPs) to be administered and for the allergen test to be conducted
4. Subjects who have decided to voluntarily participate in the study and provided a written consent regarding observance of precautions after having been informed of and having fully understood the objectives, methods, and effects of the study in detail
5. Subject with a Body Mass Index (BMI)* between 18.5 and 30.0 kg/㎡

   * BMI = Weight(kg) / Height (m)²

Exclusion Criteria:

[Medication History]

1. Subjects who were administered or treated with the following medications during the periods mentioned below from the screening visit (Visit 1) or are scheduled for administration during the study º Within one month prior to the screening visit: Hyaluronidase, Chemotherapeutic agent, Immunosuppressive agent º Within 14 days prior to the screening visit: Glucocorticoid (e.g., Dexamethasone, Prednisone, etc.), Antihistamine (e.g., Chlopheniramine, Hydroxyzine, Ketotifen, etc.) Non-steroidal anti-inflammatory drugs(NSAIDs)(e.g., Aspirin, Aceclofenac, etc.), Penicillin (e.g., Amoxicillin, Ampicillin, etc.), Cephalosporins(e.g., Cefaclor, Cefadroxil, Cefixime, etc.), Sulfa antibiotics (e.g., Sulfadiazine, Sulfamethoxazole, etc.) and Quinolones (e.g., Ciprofloxacin, Levofloxacin, etc.)

   [Medical History and Concurrent Disease]
2. Subjects with a history of anaphylaxis
3. Subjects who had an acute fever with a temperature over 37.5℃ within seven days before the expected date of administration of the IPs or had a symptom from which an acute disease is inferred within 14 days before the expected date of administration
4. Subjects with a history of drug abuse or alcoholism or subjects who are suspected of drug abuse or alcoholism before the screening visit(Visit 1)
5. Subjects with a systolic blood pressure(SBP) > 140 mmHg or < 80 mmhg or a diastolic blood pressure (DBP) > 90 mmHg or < 50 mmHg by the vital sign tests at the screening visit (Visit 1)
6. Subjects with clinically significant abnormal results by the laboratory tests, physical examinations, vital sign tests, or electrocardiography at the screening visit (Visit 1)
7. Subjects with a total protein of 5.5 g/dL or less by the blood chemistry tests at the screening visit (Visit 1)
8. Subjects determined by the investigator to be ineligible for the study due to the following serious medical or psychiatric disorders

   ① Cardiac disease : Myocardial infarction, coronary artery bypass, arrhythmia or other serious cardiac diseases, venous stasis, etc.

   ② History of malignant tumors within five years before the screening visit (Visit 1)

   ③ Immunological disorders that may affect the immunological system [e.g., Rheumatoid arthritis, Human immunodeficiency virus (HIV), Hepatitis B virus (HBV), Hepatitis C Virus (HCV), etc.]

   ④ Mental illness such as alcoholism

   ⑤ Disorders in the respiratory, hepato-biliary, nervous, endocrine, genitourinary, and musculoskeletal systems determined to be clinically significant by the investigator
9. Subjects who are allergic to the Chinese hamster ovary (CHO) proteins, bee venoms, bee venom acupuncture, bovine proteins, or ovine proteins
10. Subjects who are allergic or hypersensitive to the IPs or its ingredient

    [Others]
11. Women of child-bearing potential or in the period of less than 12 months after menopause who have been confirmed positive in the pregnancy test (Urine hCG or Serum β hCG) at the screening visit (Visit 1)
12. Breast-feeding women or women who plan to breast-feed during the study
13. Subject who plan to participate in another study or subjects who participated in another study and were administered or treated with an investigational product (or investigational device) within six months before the screening visit (Visit 1)
14. Subjects determined to be ineligible for the study by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Part I : Incidence of drug allergic reaction within 48 hours after the intradermal injection of the IPs | within 48 hours after the intradermal injection of the IPs
  Drug allergic reactions include both immediate allergic reaction (within 30 minutes after IPs administration) and delayed drug allergic reaction (between 30 minutes and 48 hours after IPs administration).
Part II : Incidence of adverse events after the subcutaneous injection of the IPs | at 30 minutes after the intradermal injection
Part II : Incidence of adverse events after the subcutaneous injection of the IPs | at 48 hours after the intradermal injection

SECONDARY OUTCOMES:
Incidence of immediate drug allergic reaction within 30 minutes after the intradermal injection of the IPs | within 30 minutes after the intradermal injection in Part I
  Immediate drug allergic reaction is defined as drug allergic reaction with a wheal of ≥8 mm with/without a pseudopod, or an erythema or localized itching at the injection site within 30 minutes after the intradermal injection of the IPs
Incidence of delayed drug allergic reaction at 30 minutes and 48 hours after the intradermal injection of the IPs | between 30 minutes and 48 hours after the intradermal injection in Part I
  Delayed drug allergic reaction is defined as drug allergic reaction occurring between 30 minutes and 48 hours after the intradermal injection of the IPs, including, but not limited to, redness, rash, wheals, edema, erythema, or acute generalized exanthematous pustulosis and erythema multiforme, etc., at the injection site
Incidence of injection site reaction at 30 minutes and 48 hours after the administration of the IPs | at 30 minutes and 48 hours after the intradermal injection
  At each time points, wheals, erythema, localized itching and others are collected as adverse events after the administration of the IPs
Size of the wheal or erythema at 30 minutes and 48 hours after the administration of the IPs | at 30 minutes and 48 hours after the intradermal injection
  At each time points, the size of a wheal or erythema is measured. To determine the size of the wheal or erythema, the long diameter and the short diameter orthogonally intersection the long diameter at the center or the long diameter are measured and the mean of the two diameters is calculated for the size of the wheal or erythema.

CONTACTS AND LOCATIONS:
Overall Officials: Beom Joon Kim, MD, Ph.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hospital, Seoul, Heukseok-ro, Dongjak-gu, South Korea